CLINICAL TRIAL: NCT00251043
Title: Antepartum Study on Use of Interpersonal Psychotherapy at 3 New York City Sites
Brief Title: Antepartum Study on Use of Interpersonal Psychotherapy at 3 New York City Site
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #4830/6040R; R01MH069915 (NIH); R01MH069915-01A2 (NIH); 4830/6040R (Other: New York State Psychiatric Institute)
Record Dates: First submitted 2005-11-07; First posted 2005-11-09 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Depression
Keywords: Pregnancy; Antepartum Depression; Major Depression
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Interpersonal Psychotherapy; Pregnancy; Psychotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will Psychotherapy weekly for 12 weeks
  Interventions: Behavioral: Interpersonal psychotherapy for depression in pregnancy
- 2 (Active Comparator): Parenting Education will include 45-minute weekly sessions for 12 week
  Interventions: Behavioral: Parenting education program (PEP)

INTERVENTIONS:
Behavioral: Interpersonal psychotherapy for depression in pregnancy — IPT-P will include 45-minute weekly sessions for 12 weeks. During sessions, participants will learn ways to address emotional stressors associated with childbirth.
  Other Names: psychotherapy
  Arms: 1
Behavioral: Parenting education program (PEP) — PEP will include 45-minute weekly sessions for 12 weeks. During sessions, participants will learn about the stages of pregnancy, childbirth, and early infant development.
  Other Names: PEP
  Arms: 2

SUMMARY:
This study will evaluate the effectiveness of interpersonal psychotherapy in treating pregnant women with depression.

DETAILED DESCRIPTION:
The prevalence of antepartum depression (APD) increases twofold in women with poor social supports, low socioeconomic status (SES), and negative life events. APD may cause low birth weight, premature labor, and eclampsia. APD is also one of the best predictors of postpartum depression (PPD), which in turn may lead to impaired emotional and cognitive development of the infant. Therefore, early treatment of APD is important for the well-being of both the woman and her infant. Forms of psychotherapy have been successful in treating depression in the general population, but more research is necessary to determine the safest and most effective means of treating depression in pregnant women. Interpersonal psychotherapy targets interpersonal events and relationships. Interpersonal psychotherapy adapted for ADP may be effective in reducing depression, preventing PPD, and improving maternal infant attachment. This study will compare the effectiveness of interpersonal psychotherapy for depression in pregnancy (IPT-P) with a parenting education program (PEP) in treating depressed pregnant women who may be affected by SES and psychosocial factors.

Participation in this single-blind study will last through 6 months postpartum. Potential participants will first undergo initial screening, which will include a 90-minute interview with a psychiatrist and a mood assessment with an independent evaluator. Eligible participants will then be randomly assigned to receive 12 weeks of either IPT-P or PEP. Participants in both groups will attend 45-minute weekly sessions prior to delivery of their babies. At each visit, participants will complete questionnaires about mood, anxiety, mother-infant bonding, and daily function. Participants receiving IPT-P will learn ways to address emotional stressors associated with childbirth and will be regularly contacted by a therapist to discuss feelings and emotions. Participants receiving PEP will learn about the stages of pregnancy, childbirth, and early infant development.

After delivery, participants will receive weekly phone calls from a therapist during the first 4 weeks. All participants will then return for five evaluation visits, occurring at Weeks 4, 8, 12, 26, and 24 postpartum. During these visits, a therapist will evaluate participants' moods and mother-infant attachment and will refer participants to treatment if needed. The first four visits will be individual evaluations and the last visit will be a group meeting with other mothers and their infants.

ELIGIBILITY:
Inclusion Criteria:

* Depressed Pregnant women between 18-45 years
* Meets diagnostic criteria for a major depressive disorder
* Reads and understands English or Spanish
* Physically healthy without serious medical illness
* Between 12 and 33 weeks gestation
* Meets diagnostic criteria of DSM-V for a major depressive disorder
* HAM-D score > 12
* EPDS>10

Exclusion Criteria:

* Drug or alcohol abuse in the 6 months prior to study entry
* Acute risk for suicide
* Clinically significant co-morbid Axis1 disorders
* High risk pregnancy or medical conditions that affect pregnancy when participation in the study will add to risk or compromise the medical condition
* History of or present non-drug induced psychosis
* Currently taking antidepressant medication
* Exclude severe (HAM-D (17 items) score >24) depression prominent vegetative symptoms and or loss of appetite

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 142 (Actual)
Dates: Start 2005-09; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Depression | Measured weekly for 12 weeks antepartum and Weeks 4, 8, 12, 16, and 24 postpartum

SECONDARY OUTCOMES:
Mother-infant bonding | Measured at Weeks 4, 8, 12, 16, and 24 postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Margaret G. Spinelli, MD, Principal Investigator — New York State Psychiatric Institute; Jean Endicott, PhD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Background] Spinelli MG, Endicott J. Controlled clinical trial of interpersonal psychotherapy versus parenting education program for depressed pregnant women. Am J Psychiatry. 2003 Mar;160(3):555-62. doi: 10.1176/appi.ajp.160.3.555. PMID 12611838
- [Derived] Spinelli MG, Endicott J, Goetz RR, Segre LS. Reanalysis of efficacy of interpersonal psychotherapy for antepartum depression versus parenting education program: initial severity of depression as a predictor of treatment outcome. J Clin Psychiatry. 2016 Apr;77(4):535-40. doi: 10.4088/JCP.15m09787. PMID 27137422
- [Derived] Spinelli MG, Endicott J, Goetz RR. Disagreement between therapist raters and independent evaluators in a controlled clinical trial of interpersonal psychotherapy for depressed pregnant women. J Psychiatr Pract. 2015 Mar;21(2):114-23. doi: 10.1097/01.pra.0000462604.79606.4e. PMID 25782762
- [Derived] Spinelli MG, Endicott J, Goetz RR. Increased breastfeeding rates in black women after a treatment intervention. Breastfeed Med. 2013 Dec;8(6):479-84. doi: 10.1089/bfm.2013.0051. Epub 2013 Aug 24. PMID 23971683
- [Derived] Spinelli MG, Endicott J, Leon AC, Goetz RR, Kalish RB, Brustman LE, Carmona YR, Meyreles Q, Vega M, Schulick JL. A controlled clinical treatment trial of interpersonal psychotherapy for depressed pregnant women at 3 New York City sites. J Clin Psychiatry. 2013 Apr;74(4):393-9. doi: 10.4088/JCP.12m07909. PMID 23656847